CLINICAL TRIAL: NCT07261631
Title: A Phase I Open-label, Multi-center Study to Evaluate the Safety, Tolerability, Dosimetry, and Preliminary Activity of [177Lu]Lu-DFC413 and Safety and Imaging Properties of [68Ga]Ga-NNS309 in Patients With Solid Tumors
Brief Title: Phase I Study of [177Lu]Lu-DFC413 in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGCJ904A12101; 2025-521702-18 (Other: EU CTIS)
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Non-Small Cell Lung Cancer; HR+/HER2- Ductal and Lobular Breast Cancer; Triple Negative Breast Cancer; Colorectal Cancer; Soft Tissue Sarcoma
Keywords: PDAC; NSCLC; Breast cancer; CRC; STS; Radioligand therapy (RLT)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Colorectal Neoplasms; Sarcoma; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients will receive 68Ga-NNS309 and only patients with tumor uptake will receive 177Lu-DFC413
  Interventions: Drug: 68Ga-NNS309; Drug: 177Lu-DFC413

INTERVENTIONS:
Drug: 68Ga-NNS309 — Diagnostic investigational radiopharmaceutical
Drug: 177Lu-DFC413 — Therapeutic investigational radiopharmaceutical

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, dosimetry and preliminary efficacy of [177Lu]Lu-DFC413 and safety and imaging properties of [68Ga]Ga-NNS309 in patients aged ≥ 18 years with solid tumors

DETAILED DESCRIPTION:
GCJ904A12101 is first-in-human (FIH), phase I, open label study that consists of a dose escalation part followed by a dose expansion part. In both parts of the study, patients will initially be imaged with a 68Ga-NNS309 positron emission tomography (PET)/ computed tomography (CT) or PET/magnetic resonance imaging (MRI) scan and will be evaluated for eligibility for 177Lu-DFC413 treatment. Patients eligible for treatment will receive 177Lu-DFC413. In the escalation part, different doses of 177Lu-DFC413 will be tested to assess its safety, tolerability, and dosimetry and identify the recommended radioactive administered dose(s) (RD(s)) for further evaluation. The expansion will include arms based on tumor type. The end of study will occur when all patients per disease group in the expansion part have completed the follow-up for disease progression or discontinued from the study for any reason, and all patients have completed treatment and the long-term follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years with one of the following indications:
* Locally advanced unresectable or metastatic PDAC, with disease progression following, or intolerance to cytotoxic therapy, unless patient was ineligible to receive such therapy
* Locally advanced unresectable or metastatic NSCLC without any actionable genomic alterations with disease progression following, or intolerance to chemotherapy and immunotherapy, unless patient was ineligible to receive such therapy, or locally advanced unresectable or metastatic NSCLC with an actionable genomic alteration with disease progression following, or intolerance to chemotherapy and targeted therapy, unless patient was ineligible to receive such therapy
* Locally advanced unresectable or metastatic HR+/HER2- ductal and lobular breast cancer with disease progression following, or intolerance to, hormone therapy and CDK inhibitor, and at least one additional line of therapy, unless patient was ineligible to receive such therapy
* Locally advanced unresectable or metastatic triple negative breast cancer (TNBC) with disease progression following, or intolerance to, at least two lines of therapy, unless patient was ineligible to receive such therapy
* Locally advanced or metastatic unresectable CRC with disease progression following, or intolerance to cytotoxic chemotherapy, unless patient was ineligible to receive such therapy. Patients with known microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) status must also have had disease progression following, or intolerance to, immune checkpoint inhibitor therapy, unless patient was ineligible to receive such therapy
* (Dose expansion only) Locally advanced unresectable or metastatic soft tissue sarcoma (excluding GIST and Kaposi) with disease progression following, or intolerance to, at least one line of systemic therapy
* Patients must have lesions showing 68Ga-NNS309 uptake

Exclusion Criteria:

* Absolute neutrophil count (ANC) < 1.5 x 109/L, hemoglobin < 9 g/dL, or platelet count < 100 x 109/L
* QT interval corrected by Fridericia's formula (QTcF) ≥ 470 msec
* eGFR < 60 mL/min, calculated using CKD-EPI 2021 or measured
* Unmanageable urinary tract obstruction or urinary incontinence
* Presence of symptomatic CNS metastases, or CNS metastases that require local CNS-directed therapy
* Any prior radioligand therapy
* Radiation therapy within 4 weeks prior to the first dose of [177Lu]Lu-DFC413

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2029-05-09 (Estimated); Study Completion 2029-05-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities of 177Lu-DFC413 | Within first treatment cycle, up to maximum 6 weeks
  A dose limiting toxicity (DLT) is defined as any adverse event or abnormal laboratory value of CTCAE (version 5.0) Grade 3 or higher that occurs within the DLT evaluation period and that is not primarily related to disease, disease progression, intercurrent illness, or concomitant medications with a few exceptions defined in the study protocol. Other clinically significant toxicities may be considered to be DLTs, even if not Grade 3 or higher.
Incidence and severity of adverse events and serious adverse events of 177Lu-DFC413 | From study treatment start up to approximately 42 months
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs) and Serious Adverse Event (TESAEs) and through the monitoring of relevant clinical and laboratory safety parameters.
Dose modifications for 177Lu-DFC413 | From study treatment start until last dose of study treatment, assessed up to approximately 24 weeks
  Dose modifications (dose interruptions and reductions) for 177Lu-DFC413 will be assessed and summarized using descriptive statistics. The number of patients with dose modification and the reasons will be summarized by treatment groups.
Dose intensity for 177Lu-DFC413 | From study treatment start until last dose of study treatment, assessed up to approximately 24 weeks
  Dose intensity for 177Lu-DFC413 will be assessed and summarized using descriptive statistics. Dose intensity is computed as the ratio of actual cumulative dose received and actual duration of exposure.

SECONDARY OUTCOMES:
Overall response rate (ORR) | From study treatment start up to 6 months
  ORR is defined as the proportion of patients with a BOR of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines.
Duration of Response (DOR) | From study treatment start up to 6 months
  DOR is the time between the first documented response (CR or PR) and the date of progression according to RECIST v1.1 guidelines, or death due to any cause.
Disease control rate (DCR) | From study treatment start up to 6 months
  DCR is defined as the proportion of patients with a BOR of CR, PR or stable disease according to RECIST v1.1 guidelines.
Progression free survival (PFS) | From study treatment start up to 6 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression according to RECIST v1.1 guidelines or death due to any cause.
Area Under the Curve (AUC) of 177Lu-DFC413 | Up to 8 days after first dose
  The 177Lu-DFC413 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. AUC will be determined by non-compartmental methods.
Total body clearance of 177Lu-DFC413 | Up to 8 days after first dose
  The 177Lu-DFC413 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Total body clearance will be determined by non-compartmental methods.
Observed maximum blood concentration (Cmax) of 177Lu-DFC413 | Up to 8 days after first dose
  The 177Lu-DFC413 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Cmax will be determined by non-compartmental methods.
Observed maximum radioactivity concentration (Rmax) of 177Lu-DFC413 | Up to 8 days after first dose
  The 177Lu-DFC413 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Rmax will be determined by non-compartmental methods.
Volume of distribution (Vz) of 177Lu-DFC413 during the terminal phase | Up to 8 days after first dose
  The 177Lu-DFC413 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. Vz will be determined by non-compartmental methods.
Terminal elimination half-life (T1/2) of 177Lu-DFC413 | Up to 8 days after first dose
  The 177Lu-DFC413 pharmacokinetic analysis will be performed based on decay-corrected blood radioactivity concentration data converted to mass units. T1/2 will be determined by non-compartmental methods.
Urinary excretion of radioactivity expressed as a percentage of injected dose (%ID) | Up to 3 days after first dose
  Urine elimination data for 177Lu-DFC413 will be assessed based on decay-corrected urine radioactivity concentration data. Urine elimination data will be expressed as percentage of injected dose (%ID).
Renal clearance of 177Lu-DFC413 | Up to 3 days after first dose
  Urine samples will be collected over specified time intervals and analyzed for radioactivity. Renal clearance of 177Lu-DCF413 will be summarized using descriptive statistics.
Absorbed dose of 177Lu-DFC413 | Up to 8 days after first dose
  Time activity curves (TACs) for the various organs and tumor lesions will be produced as fraction of injected activity per gram of tissue (%ID/g) as a function of time.
Incidence and severity of adverse events and serious adverse events of [68Ga]Ga-NNS309 | Up to 3 days after administration
  The distribution of adverse events will be done via the analysis of frequencies for TEAEs and TESAEs and through the monitoring of relevant clinical and laboratory safety parameters.
Visual and quantitative assessment of [68Ga]Ga-NNS309 uptake in normal tissues and tumor lesions over time | Up to 3 days after administration
  After [68Ga]Ga-NNS309 administration, [68Ga]Ga-NNS309 PET/CT or PET/MRI will be performed. Standardized uptake values (SUVs) of [68Ga]Ga-NNS309 in normal tissues and tumor lesions over time will be summarized.

CONTACTS AND LOCATIONS:
Locations (4):
- Novartis Investigative Site, Montreal, Quebec, Canada
- Israel (2):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Tel Aviv
- Novartis Investigative Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.